CLINICAL TRIAL: NCT06369025
Title: Improving Children's Mental Health by Preventing Teacher and Family Violence: A Pilot Cluster-randomized Controlled Trial
Brief Title: Preventing Physical and Emotional Violence by Parents and Teachers in Public Schools in Tanzania (ICC-T/ICC-P_Tanz)
Acronym: PreVio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Collaborators: Technical University of Munich (Other); Dar es Salaam University College of Edcuation (Unknown); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Tobias Hecker, PhD, Prof. Dr., Bielefeld University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PreVio
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Violence
Keywords: school violence; teacher violence; parental violence; family violence; children; public schools; primary schools

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICC-T & ICC-P (Experimental): ICC-T: 5 days with 8 hours of training for teachers. Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting.
  ICC-P: 4 days with 8 hours of training for parents. Core training components include parents-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened children and implementation of the training materials into the daily home setting
  Interventions: Behavioral: Interaction Competencies with Children
- Monitoring condition (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Interaction Competencies with Children — Interaction Competencies with Children - for Teachers (ICC-T) Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting.
  Interaction Competencies with Children - for Parents (ICC-P) Core training components include parents-child interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the home
  Arms: ICC-T & ICC-P

SUMMARY:
More than 1.7 billion children worldwide experience violence in their upbringing. Prevalence rates are particularly high in Africa. Toxic stress associated with violence impacts the developing brain. This affects behavioral, social, and emotional functioning of children. The present project will test an intervention that simultaneously aims at reducing violence against children at home and at school. Within the project, (1) the feasibility, acceptability, and cost-effectiveness of the Intervention and (2) the initial effectiveness of reducing parental and teacher violence will be tested. To this end, a mixed-methods two-arm school-based pilot cluster-randomized controlled trial (CRCT) in Tanzania will be conducted.

One unique and novel aspect of this project is to test a school-based intervention approach that targets both teachers and parents. A school-based approach including both teachers and parents has the following key advantages: (1) parents of different social, economic, and educational backgrounds can be motivated to participate and (2) using the existing infrastructure of schools reduces costs and will later improve the scalability of the program. The project is bringing together the global health, development economy, and psychological perspectives to promote our collaboration within the German global health community and with research and policy partners in Tanzania.

DETAILED DESCRIPTION:
The study is a two-arm cluster-randomized controlled trial with 16 primary schools (clusters) in the Urban District of Morogoro in Eastern Tanzania as level of randomization. The eligible schools are located in 20 wards (smallest administrative unit). To avoid cross-over effects between the study conditions, only one school per ward will be selected. To select the final sample of schools, 16 out of the 20 wards schools will be randomly selected and then one school from each ward. Then pairs of schools will be randomly formed. These has primarily logistical reasons: Due to the short project period (12 months), the implementation of the intervention will start after completion of the baseline assessment in the first pair of schools and after randomly allocation of the first school to the intervention condition. The selection and allocation of the schools will be performed by an independent researcher neither belonging to the core research team nor involved in data collection process.

At each school, 45 students in the in 5th school grade, 90 parents (45 mothers & 45 fathers = 90 parents) and 25 teacher will be recruited. Thus the final sample will comprise 720 students, 720 parent pairs (720 mothers & 720 fathers) and 400 teachers at baseline across 16 schools.

The study will have two data assessment points: baseline assessment prior to the intervention, the one follow-up assessment three months after the intervention. In addition, feasibility data will be assessed in the intervention group at the beginning and the end of the intervention. The cluster-randomized control trails will additionally be accompanied by a process evaluation.Qualitative information will be collected after intervention training of parents and teachers to complement the quantitative data.

Primary outcome measures are student-, parents- and teacher-reported physical and emotional violence by the parents or teachers in the past week. Secondary outcome measures include adult-child relationship, children's emotional and behavioral problems, quality of life, parents' and teachers' stress level and school climate.

ELIGIBILITY:
General:

Inclusion Criteria:

Schools:

* Public primary schools
* at least 45 students in selected class/ stream
* least 25 but no more than 50 employed teacher in selected school.

All participants:

- Written informed consent (if underaged by parents (written) & minors themselves (orally)

Students:

* Enrollment in selected public primary school, age between 9 and 13 years
* living with their caregiver or parents near to the schools

Teachers:

* employed at the selected schools
* aged between 18 and 60 years of age (statutory retirement age)

Parents:

* their child is participating in the study and is enrolled in a study's eligible school,
* social parent (the parent currently taking care of the child independent of the biological relationship to the children; social parents can be biological parents, step-parents, foster parents, relatives, etc.)
* aged between 16 and 80 years of age

Exclusion criteria (all participants):

* Acute drug or alcohol intoxication,
* acute psychotic disorder
* severe mental disabilities

Ages: 9 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1848 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Reduction of children's exposure to emotional and physical violence by parents and teachers | The CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess children's self-reported experiences of emotional and physical violence by parents at home and teachers at school in the past week. Higher scores indicate higher levels of violence that is used by parents or teachers. A stronger reduction of exposure to violence in the children of parents and teachers of the intervention group compared to the control group is hypothesized.
Reduction of parents' or teachers' use of emotional and physical violence | The CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess parents' and teachers' use of emotional and physical violent discipline measures against children in the past week. Higher scores indicate higher levels of violence that is used by parents or teachers. A stronger reduction of violence use by parents and teachers of the intervention group compared to the control group is hypothesized.

SECONDARY OUTCOMES:
Change of parents' and teachers' attitudes towards emotional and physical violence | The adapted version of CTS will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  Teachers' and parents' attitudes towards emotional and physical violence will be assessed with an adapted version of the Conflict Tactic Scale (CTS). Higher scores indicate higher levels of positive attitudes towards violence. A stronger reduction of favourable attitudes towards violence of parents and teachers of the intervention group compared to the control group is hypothesized.
Improvement of children's mental health | The PSC-Y will be used at T1 (baseline, prior to intervention) and T2 (first follow-up, 3 months after intervention)
  The Pediatric Symptom Checklist - Youth Report (PSC-Y) will assess children's emotional and behavioral problems reported by children and parents. Higher scores indicate higher levels of children's mental health problems. A stronger improvement of mental health problems in the children of parents and teachers of the intervention group compared to the control group is hypothesized.
Increase of children's quality of life | The KIDSCREEN-10 will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The KIDSCREEN-10 will assess children's quality of life reported by children and parents. Higher scores indicate higher levels of children's quality of life. A stronger increase of quality of life in the children of parents and teachers of the intervention group compared to the control group is hypothesized.
Improvement of school climate | The Teacher Relationship with Colleagues will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Teacher Relationship with Colleagues will assess school climate reported by teachers. Higher scores indicate higher quality of school climate. A stronger increase of school climate quality in the intervention group compared to the control group is hypothesized.

OTHER OUTCOMES:
Reduction of children's perceived stress | The Stress Scale for Kids will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Stress Scale for Kids will assess the perceived stress of children reported by children. Higher scores indicate higher levels of stress. A stronger decrease of children's perceived stress in the children of parents and teachers of the intervention group compared to the control group is hypothesized.
Reduction of parents' and teachers' perceived stress | The Parental Stress Scale and the Teachers Stress Inventory will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Parental Stress Scale will assess the perceived stress of parents reported by parents. The Teachers Stress Inventory will assess the perceived stress of teachers reported by teachers. Higher scores indicate higher levels of stress. A stronger decrease of parents' and teachers' perceived stress in the intervention group compared to the control group is hypothesized.
Improvement of teachers' decision making | Teacher Participation in Decision Making will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Teacher Participation in Decision Making will assess the teachers' decision making strategies reported by teachers. Higher scores indicate better decision making strategies. A stronger increase indecision making strategies in the intervention group compared to the control group is hypothesized.
Improvement of teachers' self-efficacy | Teachers Sense of Efficacy Scale will be used at T1 (baseline, prior to intervention) and T2 (follow-up, 3 months after intervention)
  The Teachers Sense of Efficacy Scale will assess the teachers' self-efficacy reported by teachers. Higher scores indicate higher levels of self-efficacy. A stronger increase of self-efficacy in the intervention group compared to the control group is hypothesized.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hecker, Prof. Dr., Principal Investigator — Bielefeld University
Locations (1):
- Daressalaam University College of Education, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The ICC-T intervention is being tested in various other countries including Haiti, Ghana, Tanzania and Uganda. ICC-P is being pilot tested in Tanzania. We will share anonymized data with project partners from the different countries for combined and/or comparative analyses. In addition, we will share anonymized data with other researchers working on prevention of violence against children in school settings for the purpose of conducting synthesizing analyses such as meta-analyses. Finally, the anonymized data collected in the study will be made publicly available in a data repository.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The anonymized data will be made publicly available after completion of the project in 2027
Access Criteria: open source

REFERENCES:
- [Derived] Mattonet K, Kabelege E, Mkinga G, Kolwey L, Nkuba M, Masath FB, Hermenau K, Schupp C, Steinert JI, Hecker T. School-based prevention of teacher and parental violence against children: Study protocol of a cluster-randomized controlled trial in Tanzania. BMC Public Health. 2024 Aug 31;24(1):2367. doi: 10.1186/s12889-024-19888-7. PMID 39217292